CLINICAL TRIAL: NCT02287675
Title: A Randomized, Double-Blinded Trial Comparing Lymphoseek and 99mTc-Sulfur Colloid With Regard to Pre-op Imaging and Imaging Drug Kinetics and Intra-op Lymphatic Mapping and Sentinel Lymph Node Biopsy Findings in Patients With Breast Cancer
Brief Title: Sentinel Lymph Node Biopsy Findings in Patients With Breast Cancer
Acronym: Lymphoseek
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KHNIC-P14-N001
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Sentinel Node
MeSH Terms: conditions — Breast Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lymphoseek (Active Comparator): Lymphoseek (technetium Tc 99m tilmanocept) Injection is indicated for lymphatic mapping with a hand-held gamma counter to assist in the localization of lymph nodes draining a primary tumor site in patients with breast cancer or melanoma and guiding sentinel lymph node biopsy using a hand-held gamma counter in patients with clinically node negative squamous cell carcinoma of the oral cavity.
  Interventions: Drug: Lymphoseek
- Sulfur Colloid (Active Comparator): Technetium Tc 99m Sulfur Colloid Injection is a radioactive diagnostic agent indicated for use as follows:
  In adults, to assist in the:
  * localization of lymph nodes draining a primary tumor in patients with
  * breast cancer or malignant melanoma when used with a hand-held gamma counter.
  * evaluation of peritoneovenous (LeVeen) shunt patency in adults.
  Interventions: Drug: Sulfur Colloid

INTERVENTIONS:
Drug: Lymphoseek — Subjects will receive a single intradermal injection of Lymphoseek followed by SPECT imaging conducted in two phases: initial sequential planar imaging at 30 to 60 second intervals for the first 60 minutes and repeated at 90 minutes and 120 minutes, as indicated, for identification of the SLN followed by SPECT/CT for higher resolution imaging in transaxial, coronal, and sagittal planes. Subjects will then proceed to surgery for lymphatic mapping. Lymphoseek positivity will be based upon radioactivity counts derived from the application of the handheld gamma probe ex vivo. Tumor resection or mastectomy will be performed according to standard procedures.
  Other Names: technetium Tc 99m tilmanocept
  Arms: Lymphoseek
Drug: Sulfur Colloid — Subjects will receive a single intradermal injection of 99mTc-SC followed by SPECT imaging conducted in two phases: initial sequential planar imaging at 30 to 60 second intervals for the first 60 minutes and repeated at 90 minutes and 120 minutes, as indicated, for identification of the SLN followed by SPECT/CT for higher resolution imaging in transaxial, coronal, and sagittal planes. Subjects will then proceed to surgery for lymphatic mapping. 99mTc-SC positivity will be based upon radioactivity counts derived from the application of the handheld gamma probe ex vivo. Tumor resection or mastectomy will be performed according to standard procedures.
  Other Names: 99mTc-SC; 99mTc-SC Sulfur Colloid
  Arms: Sulfur Colloid

SUMMARY:
To compare the kinetics and efficacy of two functionally different diagnostic agents, Lymphoseek (CD206 receptor targeted) and 99mTc-Sulfur Colloid (SC) (Sulfur Colloid non-specific mapping agent) in intraoperative lymphatic mapping (ILM) and Sentinel Lymph Node Biopsy (SLNB).

DETAILED DESCRIPTION:
Single center, blinded, randomized, parallel-group, comparative study of Lymphoseek and 99mTc-SC in the preoperative and intraoperative detection of lymph nodes in subjects with known breast cancer. All subjects will receive a single dose of 50 μg Lymphoseek radiolabeled with 0.5 millicurie (mCi) Tc 99m or 0.5 mCi of 99mTc-SC. Subjects may also receive up to 1 mL of vital blue dye (VBD) as a companion ILM agent. All radio-labeled agents will be administered in a single intradermal injection.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be female and 18 years of age or older.
* The subject must be a preoperative clinical Tis, T1, T2, T3, T4, as well as clinical N0 and clinical M0 breast cancer
* The subject must have a diagnosis of primary breast cancer.
* The subject must be a candidate for surgical intervention, either with lumpectomy and SLNB or with mastectomy and SLNB, as the treatment of her breast cancer.
* The subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of Grade 0 - 2
* The subject must provide written informed consent with Health Insurance Portability and Accountability Act (HIPAA) authorization before participating in the study

Exclusion Criteria:

* The subject has clinical or radiological or pathologic evidence of metastatic cancer, including any abnormal or enlarged clinical palpable lymph nodes or core biopsy/surgical biopsy/fine-needle-aspiration evidence of malignant cell within any lymph nodes.
* The subject has a known hypersensitivity to vital blue dye (VBD) in a case where vital blue dye was planned for use during SLNB.
* The subject has a positive pregnancy test or is lactating.
* The subject has had prior surgery to the indicated breast or axilla.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Kardan, MD, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulfur Colloid | Lymphoseek
Started | 22 | 18
Completed | 22 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lymphoseek | Sulfur Colloid | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 5 | 13 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: inches] | 63.97 (2.56) | 65.02 (2.33) | 64.55 (2.46)
Weight [Mean (Standard Deviation); unit: pounds] | 193.72 (38.9) | 178.23 (41.45) | 185.20 (40.57)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.33 (6.86) | 29.61 (6.66) | 31.28 (6.92)
Temperature [Mean (Standard Deviation); unit: Degrees Fahrenheit] | 98.28 (0.52) | 98.19 (0.66) | 98.23 (0.59)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 138.22 (23.51) | 138.86 (22.60) | 138.58 (22.72)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 80.61 (14.12) | 78.91 (15.37) | 79.68 (14.66)
pulse [Mean (Standard Deviation); unit: beats per minute] | 81.11 (10.86) | 78.5 (11.31) | 79.68 (11.04)
respiratory rate [Mean (Standard Deviation); unit: breaths per minute] | 15.44 (1.54) | 15.62 (2.04) | 15.54 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Injection Site Clearance for Lymphoseek and 99mTc-Sulfur Colloid (SC).
Description: The rate of injection site clearance is the time from radiotracer injection to peak SLN radioactive level. Injection clearance rates will be determined by planar SPECT imaging and by SPECT/CT. Subjects will undergo standard sequential planar imaging at 30 to 60 seconds intervals until the sentinel lymph node is seen. Once a sentinel node is located, a SPECT/CT will be performed for higher resolution imaging in transaxial, coronal, and sagittal planes.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lymphoseek | Sulfur Colloid
Number analyzed (Participants) | 18 | 22
minutes | 1.78 (0.85) | 0.045 (0.18)

2. Primary Outcome: Sentinel Lymph Node Uptake Rate
Description: SLN uptake rates will be determined by planar SPECT (single-photon emission computerized tomography) imaging and by SPECT/CT (CT-computed tomography). Gamma counts will be obtained at the injection site by standard sequential planar imaging at 30 to 60 seconds intervals until the sentinel lymph node is seen. Once a sentinel node is located, a SPECT/CT will be performed for higher resolution imaging in transaxial, coronal, and sagittal planes. Figures showing the percent of peak activity in the node versus time will be constructed for each radiopharmaceutical. The average uptake rate for each radiopharmaceutical will be computed and the following test will be conducted using a two-sample t-test at a two-sided α=0.05 (one-sided α=0.025) level of significance: H0 (null hypothesis): µLS ≤ µSC vs. HA (alternative hypothesis): µLS > µSC, (µLS is the average SLN uptake rate of Lymphoseek) (µSC is the average SLN uptake rate of 99mTc Sulfur Colloid).
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lymphoseek | Sulfur Colloid
Number analyzed (Participants) | 18 | 22
minutes | 59.28 (44.02) | 86.46 (54.15)

3. Secondary Outcome: Number of Intraoperatively Detected Sentinel Lymph Nodes (SLNs) Identified
Description: To compare the number of intraoperatively detected SLNs identified by Lymphoseek and 99mTc-SC on an agent cohort basis
Time Frame: 24 hours
Population: Lymph Nodes Removed Intraoperative
Measure: Number; unit: Lymph Nodes
Units Other Than Participants: Lymph Nodes
Arm/Group | Lymphoseek | Sulfur Colloid
Number analyzed (Participants) | 18 | 22
Number analyzed (Lymph Nodes) | 28 | 32
Lymph Nodes | 9 | 22

4. Secondary Outcome: Ratio of Intraoperative Gamma Counts
Description: To compare differences in the ratio of intraoperative counts for Lymphoseek vs 99mTc-SC for the hottest harvested axillary Sentinel Lymph Node (SLN) relative to the primary intradermal injection site.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lymphoseek | Sulfur Colloid
Number analyzed (Participants) | 18 | 22
Ratio | 0.1093 (0.0917) | 0.2621 (0.6105)

5. Secondary Outcome: Patient Pain Tolerance
Description: To compare patient pain tolerance (i.e., patient's perceived level of discomfort) at the injection site for Lymphoseek vs 99mTc-SC using Wong-Baker pain rating scale of 0-10, where the higher the score, the higher the pain level.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lymphoseek | Sulfur Colloid
Number analyzed (Participants) | 18 | 22
score on a scale | 0.5278 (0.88238) | 1.5682 (2.17286)

6. Secondary Outcome: Pathologic Assessment of the Excised Lymph Node(s)
Description: To compare pathologic assessment of the excised lymph node(s) to confirm the presence/absence of tumor metastases for Lymphoseek vs 99mTc-SC.
Time Frame: 24 hours
Population: Intraoperative Lymph Nodes extracted with presence of radiotracer
Measure: Count of Units; unit: Lymph Nodes
Units Other Than Participants: Lymph Nodes
Arm/Group | Lymphoseek | Sulfur Colloid
Number analyzed (Participants) | 18 | 22
Number analyzed (Lymph Nodes) | 9 | 22
Lymph Nodes
  Positive for tumor metastasis | 2 | 0
  Negative for tumor metastasis | 7 | 22

ADVERSE EVENTS:
Time Frame: From screening through follow-up, up to 50 days
Arm/Group | Lymphoseek | Sulfur Colloid
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 2/18 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoseek (N=18) | Sulfur Colloid (N=22)
Intermittent headaches (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT02287675/Prot_SAP_000.pdf
  • Informed Consent Form (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02287675/ICF_001.pdf